CLINICAL TRIAL: NCT01362673
Title: A Phase 1, Randomized, Subject- And Investigator Blind, Sponsor Open, Placebo Controlled, Single- And Multiple-Dose Escalation Study Of PF-04171327 In Healthy Adult Japanese And Western Subjects In Fasting And Fed Conditions
Brief Title: PK And Safety Study Of PF-04171327 In Healthy Japanese And Western Subjects In Fasting And Fed Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: A9391012
Record Dates: First submitted 2011-05-17; First posted 2011-05-30 (Estimated); Last update posted 2011-10-07 (Estimated); Status verified 2011-10

CONDITIONS: Healthy
Keywords: Phase 1; Pharmacokinetics; food effect; Healthy Japanese; rheumatoid arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — fosdagrocorat

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Single dose (Experimental)
  Interventions: Drug: PF-04171327; Drug: Placebo
- Multiple dose (Experimental)
  Interventions: Drug: PF-04171327; Drug: Placebo

INTERVENTIONS:
Drug: PF-04171327 — Oral single 5 mg dose as one 5 mg tablet
  Arms: Single dose
Drug: PF-04171327 — Oral single 10 mg dose as one 10 mg tablet
  Arms: Single dose
Drug: PF-04171327 — Oral single 30 mg dose as three 10 mg tablets
  Arms: Single dose
Drug: Placebo — Oral single dose as matching placebo
  Arms: Single dose
Drug: PF-04171327 — Oral multiple 20 mg doses as two 10 mg tablets for 12 days
  Arms: Multiple dose
Drug: Placebo — Oral multiple doses as matching placebo for 12 days
  Arms: Multiple dose

SUMMARY:
This Phase 1 study is the first clinical trial in Japanese subjects. This study is designed to evaluate the single- and multiple-dose pharmacokinetics, safety and tolerability of PF-04171327 oral tablet in healthy adult Japanese and Western subjects in fasting and fed conditions.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects of non childbearing potential between the ages of 18 and 55 years.
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >45 kg (99 lbs).
* Japanese subjects who have four Japanese grandparents born in Japan.

Exclusion Criteria:

* Confirmed fasting glucose more than 100 mg/dL at Screening and Day 0 in both Cohort A and B.
* Corticosteroid use of more than 5 mg prednisone equivalent per day for more than 6 weeks.
* Evidence or history of clinically significant hematological (including anemia), renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2011-05; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Plasma pharmacokinetic parameters for PF-00251802 : Cmax | Day 1 to Day 4 in each period of Cohort A
Plasma pharmacokinetic parameters for PF-00251802 : Tmax | Day 1 to Day 4 in each period of Cohort A
Plasma pharmacokinetic parameters for PF00251802 : AUC(0-last) | Day 1 to Day 4 in each period of Cohort A
Plasma pharmacokinetic parameters for PF-00251802 : As data permit AUC(0-inf) | Day 1 to Day 4 in each period of Cohort A
Plasma pharmacokinetic parameters for PF-00251802 : As data permit t1/2 | Day 1 to Day 4 in each period of Cohort A
Plasma pharmacokinetic parameters for N-oxide metabolite (PF-04015475): Cmax | Day 1 to Day 4 in each period of Cohort A
Plasma pharmacokinetic parameters for N-oxide metabolite (PF-04015475): Tmax | Day 1 to Day 4 in each period of Cohort A
Plasma pharmacokinetic parameters for N-oxide metabolite (PF-04015475): AUC(0-last) | Day 1 to Day 4 in each period of Cohort A
Plasma pharmacokinetic parameters for N-oxide metabolite (PF-04015475): As data permit AUC(0-inf) | Day 1 to Day 4 in each period of Cohort A
Plasma pharmacokinetic parameters for N-oxide metabolite (PF-04015475): As data permit t1/2 | Day 1 to Day 4 in each period of Cohort A
Plasma pharmacokinetic parameters for PF-00251802: Cmax for Day 1 and Day 12 | Day 1 to Day 15 in Cohort B
Plasma pharmacokinetic parameters for PF-00251802: Tmax for Day 1 and Day 12 | Day 1 to Day 15 in Cohort B
Plasma pharmacokinetic parameters for PF-00251802: AUCtau for Day 1 and Day 12 | Day 1 to Day 15 in Cohort B
Plasma pharmacokinetic parameters for PF-00251802: As data permit t1/2 for Day12 | Day 1 to Day 15 in Cohort B
Plasma pharmacokinetic parameters for PF-00251802: As data permit Rac (accumulation ratio = Day 12 AUCtau/Day 1 AUCtau) for Day12 | Day 1 to Day 15 in Cohort B
Plasma pharmacokinetic parameters for PF-00251802: Ctrough | Day 1 to Day 15 in Cohort B
Plasma pharmacokinetic parameters for N-oxide metabolite (PF-04015475): Cmax for Day 1 and Day 12 | Day 1 to Day 15 in Cohort B
Plasma pharmacokinetic parameters for N-oxide metabolite (PF-04015475): Tmax for Day 1 and Day 12 | Day 1 to Day 15 in Cohort B
Plasma pharmacokinetic parameters for N-oxide metabolite (PF-04015475): AUCtau for Day 1 and Day 12 | Day 1 to Day 15 in Cohort B
Plasma pharmacokinetic parameters for N-oxide metabolite (PF-04015475): As data permit t1/2 for Day12 | Day 1 to Day 15 in Cohort B
Plasma pharmacokinetic parameters for N-oxide metabolite (PF-04015475): As data permit Rac (accumulation ratio = Day 12 AUCtau/Day 1 AUCtau) for Day12 | Day 1 to Day 15 in Cohort B
Plasma pharmacokinetic parameters for N-oxide metabolite (PF-04015475): Ctrough | Day 1 to Day 15 in Cohort B

SECONDARY OUTCOMES:
Biomarkers for bone effects: Serum procollagen type 1 N-terminal propeptide (P1NP), serum C terminal telopeptide of type I collagen (CTX), serum osteocalcin and urine N terminal telopeptide of type I collagen (uNTX). | Day 0 to Day 15 in Cohort B
Biomarkers for carbohydrate and metabolic: Plasma cortisol, serum glucose, plasma insulin and serum adiponectin. | Day 0 to Day 15 in Cohort B

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Glendale, California, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A9391012&StudyName=PK%20And%20Safety%20Study%20Of%20PF-04171327%20In%20Healthy%20Japanese%20And%20Western%20Subjects%20In%20Fasting%20And%20Fed%20Conditions